CLINICAL TRIAL: NCT05451589
Title: Improving Physical and Psychosocial Functioning in Older Adults: A Community Health Worker-Led Intervention
Brief Title: A Trial of a Positive Psychology Intervention for Older Adults (RESET)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Detroit Department of Health (Other)
Responsible Party: Principal Investigator, Mary Janevic, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00209259; R01NR020442 (NIH)
Record Dates: First submitted 2022-07-07; First posted 2022-07-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Depressive Symptoms; Anxiety; Chronic Pain; Fatigue; Loneliness; Stress, Psychological
MeSH Terms: conditions — Depression; Anxiety Disorders; Chronic Pain; Fatigue; Stress, Psychological | interventions — Self Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESET intervention (Experimental): Participants will engage in a 7-week positive psychology and self-management group telephone-based program.
  Interventions: Behavioral: RESET
- Wellness check control (Active Comparator): Participants will receive educational information and an individual wellness check phone call from a Community Health Worker to screen for unmet social needs.
  Interventions: Behavioral: Wellness Check Control

INTERVENTIONS:
Behavioral: RESET — RESET consists of 7 weekly group phone sessions led by Community Health Workers, along with an accompanying podcast series.Topics will include positive psychology, physical activity, social connection, eating well, relaxation, and more. There will be one individual session with the Community Health Worker to screen for unmet social needs and to offer connections to resources as needed. In the group sessions, participants will set goals incorporating positive activities and strategies to improve daily functioning. Up-to-date information related to COVID-19 prevention and treatment will be provided.
  Other Names: Re-Engaging in Self-care, Enjoying Today
  Arms: RESET intervention
Behavioral: Wellness Check Control — After completing the baseline survey, control group participants will be mailed an educational packet consisting of information about COVID-19 prevention and treatment, as well as essential community resources. Control group participants will also be invited to take part in a "wellness check" telephone session with a Community Health Worker, about a half-hour long, at which a social needs screener will be administered, and any needed referrals will be made. After completing the 8-month follow up, they will have the opportunity to participate in the full intervention.
  Arms: Wellness check control

SUMMARY:
The heightened vulnerability to COVID-19 of African American older adults in Detroit, Michigan and other marginalized communities is linked to systemic racism experienced over the life course. Structural inequities also magnify the pandemic's impact on older adults' physical and psychosocial functioning. Many older adults in Detroit, burdened by poor health even before the pandemic, face a downward spiral of increased distress, reduced physical and social activity, and physical deconditioning. RESET (Re-Engaging in Self-care, Enjoying Today) is a self-management and resilience-building intervention led by community health workers (CHWs) at the Detroit Health Department (DHD). The central hypothesis of this study is that RESET, with components that include group telephone calls, a podcast series, and activity trackers, will improve psychosocial and physical functioning at 2 and 8 months. Specific aims are: 1) With input from a Community Advisory Board, modify RESET for group delivery and refine content after testing in a mini-pilot (n=10). 2) Conduct a randomized, controlled trial to assess the impact of RESET (compared to a one-time /telephone wellness check) on PROMIS-29 Psychosocial Score (a weighted combination of distress, fatigue, pain, social participation and sleep) among 456 primarily African American older adults age 50 and over who are at elevated risk of poor functioning. 3) Collect qualitative (interview) data from participants and other stakeholders, and use this data to better understand trial results, as well as to assess community impact and inform a dissemination toolkit.

ELIGIBILITY:
Inclusion Criteria:

* Any elevated physical or psychosocial symptoms as follows:

Depression: Score ≥3 on the Patient Health Questionnaire-2 (PHQ-2); Anxiety: Score >= 3 on the GAD-2 anxiety screening scale; Fatigue: Rating >=4 on a 0 to 10 scale (0 = fatigued at all and 10 = extremely fatigued); Loneliness, as indicated by a score >=6 on 3-item UCLA Loneliness Scale; Perceived stress, as indicated by a mean score >3 on the Perceived Stress Scale-4; Chronic pain: Self-reported pain in muscles or joints for >3 months, >4 (0-10 scale) mean pain intensity over last month, and >=1 day in past month when pain made it difficult to do usual activities.

* Have a cell or landline phone.
* Able to converse comfortably in English.

Exclusion Criteria:

* Serious acute illness or hospitalization in last month.
* Planned major surgery in next three months that would interfere with program participation (e.g., knee or hip replacement).
* Severe cognitive impairment or dementia.
* Any other diseases or conditions that would impair cooperation with the study team or ability to complete study procedures, as determined by the clinicians on the investigative team. This would include but not be limited to severe psychiatric disorders, active suicidal ideations or history of suicide attempts, and an uncontrolled drug and/or alcohol addiction).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS-29 Mental (Psychosocial) Summary Score | Baseline, 2 months from baseline, and 8 months from baseline
  Brief Description: The PROMIS-29 Mental (Psychosocial) Summary Score is a weighted composite of distress (depression and anxiety), pain (intensity and interference), social participation, fatigue, and sleep. Weights are provided in Hays et al (2018), "PROMIS-29 v2.0 profile physical and mental health summary scores", Quality of Life Research, 1885-1891. Scores are standardized on a T-score metric, with a mean of 50 and a standard deviation of 10 in a referent population. A higher score means more of the concept being measured.

SECONDARY OUTCOMES:
Change in PROMIS-29 Physical Summary Score | Baseline, 2 months from baseline, and 8 months from baseline
  The PROMIS-29 Physical Summary Score is a weighted composite of physical functioning (the domain weighted most heavily), pain, and social participation. Weights are provided in Hays et al (2018), "PROMIS-29 v2.0 profile physical and mental health summary scores", Quality of Life Research, 1885-1891. Scores are standardized on a T-score metric, with a mean of 50 and a standard deviation of 10 in a referent population. A higher score means more of the concept being measured.
Patient Global Impression of Change (Functioning) | 2 months from baseline, and 8 months from baseline
  How participant thinks their functioning has changed from baseline (much worse (1) to much better (7)). Higher score represents a better outcome.
Change in Connor-Davidson Resilience Scale | Baseline, 2 months from baseline, and 8 months from baseline
  This scale measures ability to bounce back from stressful times, on a 10-item scale made up of statements indicating use of resilient coping strategies, which respondents rate on a scale from (0) Never True At All to (4) True Nearly All the Time, for a total score range of 0 to 40. A higher score means greater resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT05451589/ICF_000.pdf